CLINICAL TRIAL: NCT00393874
Title: Efficacy of Adjunct Sleep Interventions for PTSD
Brief Title: Efficacy of Sleep Interventions for Posttraumatic Stress Disorder (PTSD)
Acronym: EASI-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anne Germain, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR054093; W81XWH-06-1-0257
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Anxiety Disorders; Mood Disorders; Insomnia; Nightmares
Keywords: Anxiety D/O; Mood D/O
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Sleep Initiation and Maintenance Disorders | interventions — Behavior Therapy; Prazosin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medication (Active Comparator): Treatment will be conducted under double blind conditions and will last a total of 8 weeks. Participants will also receive printed educational material about sleep hygiene developed by the American Academy of Sleep Medicine. Items include going to bed when drowsy, avoiding clock watching while awake in bed, avoidance of caffeine and alcohol, engaging in moderate exercise, and ensuring comfortable sleep environment. Clinical ratings will be obtained weekly throughout the trial.Medications will be administered in a single dose to be taken 30 minutes prior to bedtime because the onset of action occurs within 30 to 90 minutes after a single dose. The research pharmacy will prepare each dose in identical gelatin capsules to prevent identification.
  Interventions: Drug: Prazosin
- Behavioral (Active Comparator): Participants randomized to BSI will receive the intervention aimed at reducing nightmares, insomnia, and sleep avoidance behavior. The treatment will be administered over 8 weeks. The intervention sessions will consist of two individual, 45-minute treatment sessions, delivered on Weeks 1 and 3. A 45-minute "booster" session will be conducted on Week 5. Thirty-minute face-to-face contacts will be scheduled on other weeks (i.e., Weeks 2, 4, 6, 7 and 8) to address any difficulty with the treatment instructions and techniques, to answer questions that may have occurred, and to complete weekly clinical ratings (CGI-I/SR and ASES).
  Interventions: Behavioral: Behavioral Sleep Intervention
- Placebo (Placebo Comparator): Participants randomized to PLA will take 4 capsules each night, and capsule will be identical to prazosin capsules. As for participants randomly assigned to PRZ, they will receive a one-week medication supplies in daily dose dispensers. Similarly, participants will also be instructed to be ready for bed at the time they take the medication, and not to engage in any activities that will prevent them from going to bed. A placebo pill condition is included for several reasons. First, there is no approved treatment approach currently recognized as being effective for sleep disturbances associated with combat-related PTSD, and which is being withheld from subjects assigned to the placebo arm of the study. We will monitor subjects carefully and on a weekly basis.
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Behavioral Sleep Intervention — Participants will receive a workbook with information related to the intervention. The three core components are presented and discussed during these sessions are:1) education about sleep and nightmares; 2) imagery rehearsal; 3) stimulus control and sleep restriction. Session 1 focuses on education on PDSD-related insomnia, nightmares, and sleep avoidance behaviors. The rationale for imagery rehearsal will then be presented, and the technique will be practiced once. Strategies for managing intrusive thoughts and images during the practice of imagery rehearsal will be discussed. Participants will be instructed to practice this technique at least three times each day for the duration of the treatment phase. During the second 45-minute session (Week 3), sleep schedules extracted from the pre-intervention sleep diary will be used to identify goals to reduce insomnia, i.e., for sleep restricted schedules, and activities to be performed out of bed when awake.
  Other Names: Behavioral Intervention for Insomnia and Nightmares
  Arms: Behavioral
Drug: Prazosin — Participants randomized to PRZ will take 4 capsules each night (PRZ dose complemented with placebo capsules ). The target dose of prazosin is 10 mg. Some individuals may require doses up to 15 mg, (Murray Raskind, M.D., personal communication, February 4, 2005). Prazosin will be administered in an initial oral dose of 1 mg (Week 1), with titration to a maximum of 15 mg. The first increment will be of 1 mg (Week 2: 2 mg), and subsequent weekly increments according to the following schedule: Week 3: 4 mg; Week 4: 6 mg; Week 5: 10 mg; Week 6: 15 mg; Week 7: 15 mg; Week 8: 15 mg. A maximum dose of 15 mg may be necessary. Medication will be administered in a single dose to be taken 30 minutes prior to bedtime because the onset of action occurs within 30 to 90 minutes after a single dose.
  Other Names: MINIPRESS®; Vasoflex®; Hypovase®,
  Arms: Medication
Drug: Placebo — Participants randomized to PLA will take 4 capsules each night for eight weeks, all capsules will be identical to prazosin capsules. As for participants randomly assigned to PRZ, they will receive a one-week medication supplies in daily dose dispensers. Similarly, participants will also be instructed to be ready for bed at the time they take the medication, and not to engage in any activities that will prevent them from going to bed.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this research study is to evaluate and compare the effects of experimental treatments aimed at improving insomnia and nightmares in men and women military veterans between the ages of 18 and 60 years old, and who have a condition called Posttraumatic Stress Disorder. Insomnia refers to difficulty falling or staying asleep, although enough time is allowed for sleeping. Insomnia is also associated with daytime consequences, such as lack of energy, irritability, and difficulty concentrating. Nightmares are bad dreams that may or may not awaken the sleeper, and that cause discomfort during the daytime.

Chronic Posttraumatic Stress Disorder (PTSD) refers to symptoms that occur after someone experienced or witnessed a life-threatening event, and that persist for three months or more after the event. Symptoms include flashbacks, nightmares, feelings of detachment from others, sleep disturbances, irritability, anxiety, and efforts to avoid people and places associated with the life-threatening event. These symptoms occur after a life-threatening event. Symptoms that persist for more than one month indicate the presence of PTSD. In the present study, we will study people with chronic PTSD, which refers to PTSD symptoms that persist for more than 3 months.

Efficacy of a treatment is defined as the capacity to produce the desired effects. In this study, we will evaluate and compare the capacity of two active experimental treatments to reduce insomnia and nightmares associated with PTSD, and one inactive intervention, called a placebo, for people who continue to have sleep difficulties despite receiving treatment with an antidepressant medication called a selective serotonin reuptake inhibitor (SSRI, like Prozac, Paxil, Zoloft, Celexa). The two active experimental treatments are a medication, prazosin, and a brief behavioral intervention, which involves exercises and techniques to reduce nightmares and improve sleep quality. Prazosin is an approved medication by the Food and Drug Administration (FDA) against high blood pressure, but is not FDA-approved for posttraumatic insomnia and nightmares.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a prevalent disorder in military samples associated with adverse emotional and health impacts and enormous health care costs, and it is often resistant to treatment. Identification of PTSD-related factors that contribute to poor clinical and health outcomes is imperative to refine treatment strategies. Post deployment -related sleep disturbances constitute one of the factors that contribute to poor clinical and health outcomes. PTSD symptoms persist during sleep, but little clinical attention is typically devoted to nighttime symptoms. Other deployment related stress reactions are associated with sleep disturbances. Sleep disturbances are resistant to traditional PTSD treatments. There is emerging evidence that adjunct sleep-focused interventions (pharmacological or behavioral) are associated with improvements in sleep, daytime symptomatology, general emotional well being, and functioning. Therefore, sleep focused interventions may enhance treatment response and clinical outcomes in individuals exposed to trauma with consequent sleep disturbances. However, the efficacy and durability of adjunct sleep interventions have not been formally evaluated and compared. In this study, we aim at comparing the efficacy and durability of interventions targeting sleep disturbances that occurred in relation to military service and or military deployment.

The overarching objective of this study is to investigate and compare the efficacy and durability of adjunct sleep-focused interventions on sleep, daytime PTSD symptomatology, and mood in a sample of 90 male and female veterans who experience nightmares and insomnia. The specific aims and hypotheses are: 1. To investigate the efficacy of prazosin, integrated behavioral sleep intervention (IBSI), and placebo (PLA) on post deployment-related sleep disturbances; 2. To compare the efficacy of pharmacological and behavioral interventions adjunct sleep focused interventions; 3. To evaluate and compare the durability of active sleep-focused interventions on sleep, daytime PTSD symptoms, mood, and anxiety by conducting a naturalistic follow-up assessment 4 months after the end-of-treatment assessment. A secondary aim is to identify demographic, psychosocial, and clinical predictors of sleep treatment response in military veterans.

Participants will be recruited from the Pittsburgh VA Health Care System clinics and services. Treatments will be administered over an eight-week period for all conditions. Primary outcome measures include (1) Sleep Quality as determined by polysomnographic (sleep) recordings, and global scores on the Pittsburgh Sleep Quality Index (PSQI) and PSQI Addendum for PTSD (PSQI-A). Sleep response will be defined as a sleep latency < 30 minutes, and wake time after sleep onset < 30 minutes, and a sleep efficiency > 85% as determined by sleep diaries and in-home sleep studies, or a decrease in > 5 points on the Pittsburgh Sleep Quality Index. Secondary outcome measures include PTSD symptom severity as determined by the Clinician-Administered PTSD scale, Part 2, and the self-report PTSD Symptom Checklist-Military version; depression severity (as determined by the Beck Depression Inventory) anxiety (Beck Anxiety Inventory), (4) health-related quality of life (SF-36). A naturalistic follow-up assessment will be conducted four months post-treatment.

The proposed study will contribute to the development of effective therapeutic strategies for PTSD. This study will provide novel information regarding predictors of sleep treatment response in PTSD, which will contribute to facilitating care management in PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Military veterans
* Age between 18 and 55 years old
* Reports of insomnia and nightmares
* Current diagnosis of PTSD
* Currently treated with an SSRI.
* Medications and dosages will remain unchanged for the duration of the study
* Participants will agree to remain in ongoing counseling services they may be receiving prior to study entry.
* Able to read and write English
* Provision of written informed consent

Exclusion Criteria:

* Current, severe, untreated Major Depressive Disorder
* Current history of suicidality requiring hospitalization
* Current history (past 6 months) of substance or alcohol abuse
* Currently actively psychotic or bipolar disorder (past year)
* Resting blood pressure < 90/60 at the screening physical examination
* Heart rate > 100 beats/minutes
* Use of an alpha-1 antagonist agent or beta-blocker
* Refusal to follow the safety measures
* Unexpected, untreated, or serious EKG findings
* Medications and/or dosage changed in the past two months
* Unstable medical condition
* Pregnant or breast-feeding women
* Apnea-hypopnea index (AHI) > 15
* Refusal to provide information relevant to selection criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Germain, Ph.D., Principal Investigator — Department of Psychiatry University of Pittsburgh School of Medicine
Locations (1):
- Western Phychiatric Institute and Clinic, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Germain A, Richardson R, Moul DE, Mammen O, Haas G, Forman SD, Rode N, Begley A, Nofzinger EA. Placebo-controlled comparison of prazosin and cognitive-behavioral treatments for sleep disturbances in US Military Veterans. J Psychosom Res. 2012 Feb;72(2):89-96. doi: 10.1016/j.jpsychores.2011.11.010. Epub 2011 Dec 20. PMID 22281448

RESULTS

PARTICIPANT FLOW:
Groups:
- Medication: Treatment will be conducted under double blind conditions and will last a total of 8 weeks. Participants will also receive printed educational material about sleep hygiene developed by the American Academy of Sleep Medicine. Clinical ratings will be obtained weekly throughout the trial.Medications will be administered in a single dose to be taken 30 minutes prior to bedtime because the onset of action occurs within 30 to 90 minutes after a single dose.
  Participants randomized to PRZ will take 4 capsules each night (PRZ dose complemented with placebo capsules ). Prazosin will be administered in an initial oral dose of 1 mg (Week 1), with titration to a maximum of 15 mg. The first increment will be of 1 mg (Week 2: 2 mg), and subsequent weekly increments according to the following schedule: Week 3: 4 mg; Week 4: 6 mg; Week 5: 10 mg; Week 6: 15 mg; Week 7: 15 mg; Week 8: 15 mg. A maximum dose of 15 mg may be necessary.
- Behavioral: Participants randomized to BSI will receive the intervention aimed at reducing nightmares, insomnia, and sleep avoidance behavior. The treatment will be administered over 8 weeks. The intervention sessions will consist of two individual, 45-minute treatment sessions, delivered on Weeks 1 and 3. A 45-minute "booster" session will be conducted on Week 5. Thirty-minute face-to-face contacts will be scheduled on other weeks (i.e., Weeks 2, 4, 6, 7 and 8) to address any difficulty with the treatment instructions and techniques, to answer questions that may have occurred, and to complete weekly clinical ratings (CGI-I/SR and ASES).
  Participants will receive a workbook with information related to the intervention. The three core components are presented and discussed during these sessions are:1) education about sleep and nightmares; 2) imagery rehearsal; 3) stimulus control and sleep restriction.
- Placebo: Participants randomized to PLA will take 4 capsules each night, and capsule will be identical to prazosin capsules. They will receive a one-week medication supplies in daily dose dispensers. Similarly, participants will also be instructed to be ready for bed at the time they take the medication, and not to engage in any activities that will prevent them from going to bed. We will monitor subjects carefully and on a weekly basis.
  Participants randomized to PLA will take 4 capsules each night for eight weeks, all capsules will be identical to prazosin capsules. As for participants randomly assigned to PRZ, they will receive a one-week medication supplies in daily dose dispensers. Similarly, participants will also be instructed to be ready for bed at the time they take the medication, and not to engage in any activities that will prevent them from going to bed.
Period: Overall Study
Arm/Group | Medication | Behavioral | Placebo
Started | 18 | 17 | 15
Completed | 15 | 13 | 13
Not Completed | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medication | Behavioral | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 15 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (11.9) | 40.0 (14.1) | 43.6 (14.0) | 41.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 5
  Male | 16 | 14 | 15 | 45
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 15 | 50

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index
Description: Self-report measures of insomnia severity. Scores range from 0 to 28, with higher scores indicated more severe insomnia. A score < 8 is considered to reflect no significant insomnia.
Time Frame: Screening, Post, and Follow-up
Population: For the medication arm, 18 participants completed ISI at screening, 15 at post, and 12 at follow-up. For the Behavioral arm, 17 participants completed ISI at screening, 13 at post, and 12 at follow-up. For the placebo arm, 15 participants completed ISI at screening, 13 at post, and 11 at follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication | Behavioral | Placebo
Number analyzed (Participants) | 18 | 17 | 15
units on a scale
  Screening | 16.4 (4.4) | 16.5 (4.0) | 14.8 (3.7)
  Post | 9.3 (7.2) | 6.8 (5.0) | 11.8 (5.0)
  Follow-up | 7.0 (4.7) | 5.5 (5.0) | 8.7 (5.1)

2. Primary Outcome: Sleep Diary Measures
Description: Sleep diary SE, nightmare frequency Sleep diary sleep efficiency can range from 0 to 100%, and typically varies between 50% and 95%. Higher % values reflect greater sleep consolidation, i.e., greater ratio of time asleep/time in bed.
  Nightmare frequency varies between 0 and no upper limit is provided. Greater frequency of nightmares reflects greater nightmare severity.
Time Frame: baseline and post
Population: For the medication arm, 15 participants completed the sleep diary (SD) at baseline and 13 returned a SD post treatment. For the Behavioral arm, 15 participants completed the SD at baseline, and 12 returned it at follow-up. For the placebo arm, 12 participants completed the diary at baseline and 10 returned one at follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication | Behavioral | Placebo
Number analyzed (Participants) | 18 | 15 | 13
units on a scale
  SE Pre Treatment | 84.5 (11.8) | 85.5 (9.8) | 85.8 (8.0)
  SE Post Treatment | 92.2 (4.3) | 94.8 (3.0) | 90.1 (5.2)
  NF Pre Treatment | 1.0 (1.1) | .09 (1.4) | .4 (1.1)
  NF Post Treatment | .3 (.8) | .0 (.0) | .5 (1.1)

3. Primary Outcome: PSG Composite Measure
Description: Sleep Efficiency (SE) is the ratio of total time spent asleep over total time spent in bed.
  For PSG studies, (SE) typically vary between 50% and 95%. Greater values indicated more consolidated sleep.
Time Frame: Baseline sleep study and post sleep study
Population: For the medication arm, 18 participants completed a PSG study at baseline and 13 completed a PSG post treatment. For the Behavioral arm, 17 participants completed a PSG at baseline and 12 completed a PSG post-treatment. For the placebo arm, 15 participants completed a PSG at baseline and 12 completed a PSG post-treatment.
Measure: Mean (Standard Deviation); unit: percentage of time asleep vs time in bed
Arm/Group | Medication | Behavioral | Placebo
Number analyzed (Participants) | 18 | 17 | 15
percentage of time asleep vs time in bed
  Sleep Efficiency : Baseline | 82.0 (11.4) | 78.9 (2.1) | 87.1 (8.1)
  Sleep Efficiency: Post | 89.2 (7.1) | 84.5 (6.5) | 89.1 (5.0)

4. Primary Outcome: PSQI
Description: Self-report sleep quality measure. Scores range between 0 and 21, with higher scores reflecting poor sleep quality.
  A score of < or = to 5 reflects good sleep quality.
Time Frame: Baseline, post, 4 months post-treatment
Population: For the medication arm, 18 participants completed PSQI at screening, 14 at post, and 12 at follow-up. For the Behavioral arm, 17 participants completed ISI at screening, 13 at post, and 12 at follow-up. For the placebo arm, 15 participants completed ISI at screening, 13 at post, and 11 at follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Medication: Treatment will be conducted under double blind conditions and will last a total of 8 weeks. Participants will also receive printed educational material about sleep hygiene developed by the American Academy of Sleep Medicine. Items include going to bed when drowsy, avoiding clock watching while awake in bed, avoidance of caffeine and alcohol, engaging in moderate exercise, and ensuring comfortable sleep environment. Clinical ratings will be obtained weekly throughout the trial.Medications will be administered in a single dose to be taken 30 minutes prior to bedtime because the onset of action occurs within 30 to 90 minutes after a single dose. The research pharmacy will prepare each dose in identical gelatin capsules to prevent identification.
  Prazosin: Participants randomized to PRZ will take 4 capsules each night (PRZ dose complemented with placebo capsules ). The target dose of prazosin is 10 mg. Some individuals may require doses up to 15 mg, (Murray Raskind, M.D., personal
- Behavioral: Participants randomized to BSI receive the intervention aimed at reducing nightmares, insomnia, and sleep avoidance behavior. The treatment will be administered over 8 weeks. The intervention sessions will consist of two individual, 45-minute treatment sessions, delivered on Weeks 1 and 3. A 45-minute "booster" session will be conducted on Week 5. Thirty-minute face-to-face contacts will be scheduled on other weeks (i.e., Weeks 2, 4, 6, 7 and 8) to address any difficulty with the treatment instructions and techniques, to answer questions that may have occurred, and to complete weekly clinical ratings (CGI-I/SR and ASES).
  Behavioral Sleep Intervention: Participants will receive a workbook with information related to the intervention. The three core components are presented and discussed during these sessions are:1) education about sleep and nightmares; 2) imagery rehearsal; 3) stimulus control and sleep restriction. Session 1 focuses on education on PDSD-related insomnia, ni
- Placebo: Participants randomized to PLA take 4 capsules each night, and capsule will be identical to prazosin capsules. As for participants randomly assigned to PRZ, they will receive a one-week medication supplies in daily dose dispensers. Similarly, participants will also be instructed to be ready for bed at the time they take the medication, and not to engage in any activities that will prevent them from going to bed. A placebo pill condition is included for several reasons. First, there is no approved treatment approach currently recognized as being effective for sleep disturbances associated with combat-related PTSD, and which is being withheld from subjects assigned to the placebo arm of the study. We will monitor subjects carefully and on a weekly basis.
  Placebo: Participants randomized to PLA will take 4 capsules each night for eight weeks, all capsules will be identical to prazosin capsules. As for participants randomly assigned to PRZ, they will receive a one-week medicat
Arm/Group | Medication | Behavioral | Placebo
Number analyzed (Participants) | 18 | 17 | 15
units on a scale
  PSQI: Baseline | 16.4 (4.4) | 16.5 (4.0) | 14.8 (3.7)
  PSQI: Post | 7.6 (2.9) | 5.5 (3.2) | 8.9 (3.4)
  PSQI: 4-month follow up | 5.9 (2.2) | 5.5 (4.1) | 7.5 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse events and side effects were monitored throughout the duration of study participation.
Description: Events reported are (expected) side effects that were monitored throughout the duration of study participation.
  Side effects were assessed using the Asberg Side Effects Scale.
Groups:
- Medication: Treatment will be conducted under double blind conditions and will last a total of 8 weeks. Participants will also receive printed educational material about sleep hygiene developed by the American Academy of Sleep Medicine. Items include going to bed when drowsy, avoiding clock watching while awake in bed, avoidance of caffeine and alcohol, engaging in moderate exercise, and ensuring comfortable sleep environment. Clinical ratings will be obtained weekly throughout the trial.Medications will be administered in a single dose to be taken 30 minutes prior to bedtime because the onset of action occurs within 30 to 90 minutes after a single dose. The research pharmacy will prepare each dose in identical gelatin capsules to prevent identification.
  Prazosin: Participants randomized to PRZ took 4 capsules each night (PRZ dose complemented with placebo capsules ). The target dose of prazosin was 10 mg. Some individuals required doses up to 15 mg.
- Behavioral: Participants randomized to BSI received the intervention aimed at reducing nightmares, insomnia, and sleep avoidance behavior. The treatment was administered over 8 weeks. The intervention sessions consisted of two individual, 45-minute treatment sessions, delivered on Weeks 1 and 3. A 45-minute "booster" session was conducted on Week 5. Thirty-minute face-to-face contacts were scheduled on other weeks (i.e., Weeks 2, 4, 6, 7 and 8) to address any difficulty with the treatment instructions and techniques, to answer questions that had occurred, and to complete weekly clinical ratings (CGI-I/SR and ASES).
  Behavioral Sleep Intervention: Participants will receive a workbook with information related to the intervention. The three core components are presented and discussed during these sessions are:1) education about sleep and nightmares; 2) imagery rehearsal; 3) stimulus control and sleep restriction. Session 1 focuses on education on PDSD-related insomnia, ni
- Placebo: Participants randomized to PLA will take 4 capsules each night, and capsule will be identical to prazosin capsules. As for participants randomly assigned to PRZ, they will receive a one-week medication supplies in daily dose dispensers. Similarly, participants will also be instructed to be ready for bed at the time they take the medication, and not to engage in any activities that will prevent them from going to bed. A placebo pill condition is included for several reasons. First, there is no approved treatment approach currently recognized as being effective for sleep disturbances associated with combat-related PTSD, and which is being withheld from subjects assigned to the placebo arm of the study. We will monitor subjects carefully and on a weekly basis.
  Placebo: Participants randomized to PLA took 4 capsules each night for eight weeks, all capsules were identical to prazosin capsules. They received a one-week medication.
Arm/Group | Medication | Behavioral | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/15 | 3/13 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication (N=15) | Behavioral (N=13) | Placebo (N=13)
Headache, drowsiness (Nervous system disorders) | 4 (4) | 3 (3) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No